CLINICAL TRIAL: NCT03815019
Title: iKanEat: A Randomized-controlled, Multi-center Trial of Megestrol for Chronic Oral Food Refusal in Children 9 Months to 9 Years 0 Months of Age
Brief Title: iKanEat: A Randomized-controlled, Multi-center Trial of Megestrol for Chronic Oral Food Refusal in Children
Acronym: iKanEat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Ann Davis, PhD, MPH, ABPP, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00142352
Record Dates: First submitted 2019-01-17; First posted 2019-01-24 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Feeding Behavior; Feeding Disorder of Infancy or Early Childhood
Keywords: Gastrostomy Tube; G-Tube; Oral Food Refusal; Behavioral Intervention; Megestrol; Transition to Oral Feedings; Weaning
MeSH Terms: conditions — Feeding Behavior | interventions — Megestrol Acetate; Megestrol

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, placebo-controlled, double-blind clinical trial. The primary focus of the study is the evaluation of the effectiveness of treatment with megestrol as part of a 24 week behavioral feeding protocol in transitioning from tube to oral feedings in a pediatric population. Approximately 60 pediatric subjects matching the criteria for eligibility will be enrolled in the study and randomized to receive either megestrol (n=30) or placebo (n=30).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The drug will be dispensed by the investigational pharmacy at each site, who will be the only unblinded part of the team. They will receive the random codes prepared by the study statistician, and will dispense placebo/megestrol as appropriate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Megestrol (Experimental): Megestrol is a steroid and progestational drug FDA approved for treating anorexia or weight loss in patients with acquired immunodeficiency syndrome. Its use in the current protocol is "off label" to stimulate appetite in tube-fed infants and toddlers who are weaning from tube feedings and learning to eat. The precise mechanism of action that leads to increased appetite and weight gain is unknown, but is probably related to megestrol's glucocorticoid effect.
  The proposed study will use megestrol 6 mg/kg/day in two doses because this dose has been effective and safe in two previous studies using megestrol to stimulate appetite in children transitioning from tube to oral feedings. The megestrol will be dosed at full dose weeks 10-11, at 66% dose week 12, at 33% dose week 14, and fully tapered at the end of week 14. Megestrol is absorbed from the small bowel, so feeding it through the tube will be acceptable.
  Interventions: Drug: Megestrol Acetate; Behavioral: iKanEat Behavioral Intervention
- Placebo (Placebo Comparator): Subjects randomized to the placebo protocol will receive a placebo syrup identical in taste and smell to megestrol at the same intervals as those in the megestrol group but the syrup will contain no active ingredients.
  Interventions: Behavioral: iKanEat Behavioral Intervention

INTERVENTIONS:
Drug: Megestrol Acetate — The proposed study will use megestrol 6 mg/kg/day in two doses because this dose has been effective and safe in two previous studies using megestrol to stimulate appetite in children transitioning from tube to oral feedings. The megestrol will be dosed at full dose weeks 10-11, at 66% dose week 12, at 33% dose week 14, and fully tapered at the end of week 14. Megestrol is absorbed from the small bowel, so feeding it through the tube will be acceptable.
  Other Names: Megace; Megestrol
  Arms: Megestrol
Behavioral: iKanEat Behavioral Intervention — The 24 week iKanEat intervention is composed of 4 clinic visits and a series of 12 tele-visits. All visits (clinic and tele-visits) will focus directly on the oral-motor and behavioral skills necessary for oral eating.
  Tele-visits will begin by building rapport and asking for a summary of all relevant information since the last point of contact, including parent perception of changes in weight, feeding habits, progress, stress of parent/child, and illness. The majority of the time left in the 30 minute session will be spent dealing with parent concerns, which our previous project indicates may include questions about measures, questions about implementation of the iKanEat protocol, and ensuring that children/families adhere to the oral-motor and behavioral guidelines for feeding.

SUMMARY:
This is a multi-center, randomized, placebo-controlled, double-blind clinical trial. The primary focus of the study is the evaluation of the effectiveness of treatment with megestrol as part of a 24 week behavioral feeding protocol in transitioning from tube to oral feedings in a pediatric population. Approximately 60 pediatric subjects matching the criteria for eligibility will be enrolled in the study and randomized to receive either megestrol (n=30) or placebo (n=30).

DETAILED DESCRIPTION:
The primary aim of the current study is to conduct a randomized controlled trial of a 4-week course of megestrol, the only remaining medication that is part of the iKanEat protocol, to ensure that the addition of megestrol results in improved child outcomes. The second aim is to assess the safety of megestrol as part of the iKanEat protocol. Our previous work (as well as work by others) suggests that a 6 week course of megestrol can lead to adrenal insufficiency in some children, so as part of the current protocol, the investigators will assess the safety of a 4 week course of this drug.

Finally, parents of tube fed children encounter multiple psychosocial stressors regarding tube feeding. These include concerns about their child's survival due to their underlying medical issues, feelings of "failure" due to their inability to feed their child orally, increased feelings of stress around the tube feeding and decreased support from others due to the tube feeding. Our research indicates that quality of life can be poor in tube fed children, even more so than children with cancer or burns. Given the significance of these issues, the third aim of the study is to examine the effect of the transition from tube to oral feeding on parent stress and parent and child quality of life.

Aim 1: To assess the efficacy of megestrol as part of the 24 week iKanEat protocol.

Hypothesis 1: Children randomized to the megestrol group will be significantly more successful in making the transition to oral feeding (defined as obtaining at least 90% of calories orally) than children randomized to the placebo group.

Aim 2: To assess the safety of 4 weeks of megestrol as part of the 24 week iKanEat protocol.

Hypothesis 2A: Children randomized to the megestrol group will not differ from control children in morning cortisol classification level (low, average, high) and will remain within the normal range at all time points. Analyses 2B: Exploratory analysis will determine which, if any, covariates (gender, age, and diagnoses at week 0, diagnoses at birth) are related to abnormal morning cortisol levels.

Aim 3: To examine the effect of the transition from tube to oral feeding on parent stress and parent and child quality of life. Hypothesis 3A: The transition to oral feeding will temporarily increase parent stress at week 14 at the cessation of tube feeding, with a return to baseline by week 24. Hypothesis 3B: The transition to oral feeding will increase parent/child quality of life at 24 weeks compared to week 0. Children with feeding tubes have few options for treatment other than extensive inpatient stays and expensive day treatment programs. iKanEat offers an outpatient, less intensive, empirically supported effective treatment option that can improve the lives of children and families. It is imperative that the investigators determine the efficacy and safety of the protocol including 4 weeks of megestrol before the investigators move toward broad dissemination of the iKanEat protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 9 months to 9y0m at the time of consent.
2. Able to obtain parental or legal guardian written informed consent from subjects as applicable by local laws and regulations.
3. Subjects must have a G or G/J tube.
4. Subjects must receive over 80% of their total daily calorie needs from a tube in order to be classified as tube dependent.
5. Subjects must have a ≥ 3 month history of feeding problems as identified by a diagnosis from a multidisciplinary feeding team, and must have permission from the physician on the team to ensure that they are medically stable enough to participate in a weaning study.
6. Subjects must possess the oral motor skills necessary for eating. Subjects must possess behavioral skills necessary for mealtimes.

Exclusion Criteria:

1. Children receiving oral or inhaled steroids.
2. Parent has a known developmental delay or cognitive impairment that may make participation in the study difficult (children with these issues will not be excluded).
3. Children receiving intensive (defined as more than one session per month) behavioral feeding therapy with a licensed psychologist (previous behavioral feeding therapy is not an exclusion criterion; neither is current oral-motor, sensory, or speech therapy).
4. Children of non-English speaking parents.

Ages: 9 Months to 108 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Rady Children's Hospital - San Diego, San Diego, California
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards S, Hyman PE, Mousa H, Bruce A, Cocjin J, Dean K, Fleming K, Romine RS, Davis AM. iKanEat: protocol for a randomized controlled trial of megestrol as a component of a pediatric tube weaning protocol. Trials. 2021 Feb 27;22(1):169. doi: 10.1186/s13063-021-05131-w. PMID 33640012

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Megestrol | Placebo
Started | 36 | 34
Completed | 30 | 26
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Megestrol | Placebo | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.06 (2.08) | 4.20 (2.54) | 4.15 (2.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 21 | 14 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 30 | 30 | 60
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2
% calories from oral intake [Mean (Standard Deviation); unit: % calories from oral intake] | 18.51 (16.39) | 20.50 (15.43) | 19.48 (15.85)

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Transitioned to Oral Feeding
Description: The efficacy of megestrol as part of the 24 week iKanEat protocol will be measured by participants who successfully transitioned to oral feeding, defined at at least 90% calories consumed orally.
Time Frame: Weeks 0 to 24
Measure: Number; unit: Participants
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 30 | 26
Participants | 23 | 24
Statistical Analysis 1: Comparison: Megestrol; Analysis conducted using Generalized Linear Mixed Models with a logit link within SAS Proc GLIMMIX to model the binary outcome of transitioned to oral feeding (y/n) defined as at least 90 percent of calories consumed orally. Fixed effects (dummy variables) will be entered for each site as described by McNeish and Stapleton (2016) to account for the clustering of the participants within sites. This will result in essentially, a logistic regression model with appropriate standard errors; Test type: Superiority; Odds Ratio, log = 7.2218, Standard Error of Mean 13083 — Participants in the megestrol group who successfully transitioned to oral feeding
Statistical Analysis 2: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Odds Ratio, log = 9.1544, Standard Error of Mean 13083 — Participants in the placebo group who successfully transitioned to oral feeding

2. Secondary Outcome: Number of Participants With Adrenal Insufficiency as Measured by Morning Cortisol Lab Value
Description: The investigators will determine whether any of our participants in either group have adrenal sufficiency levels outside of the normal range at any time point. Should any participant have levels outside of the normal range, the investigators will descriptively examine the individual characteristics associated with this, including group assignment, medical diagnoses, sex, and age at initiation. These characteristics will be reported descriptively.
Time Frame: 10 to 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 31 | 26
Participants | 1 | 0

3. Secondary Outcome: Change in Child Quality of Life as Measured by the Infant Toddler Quality of Life Scale (ITQOL47) - Global Behavior (GB2) Subscale
Description: The investigators will model child quality of life from Week 0 to Week 24 of the intervention. The Infant Toddler Quality of Life Questionnaire™ (ITQOL) was developed for use in infants and toddlers from 2-months-to-5 years of age. The Infant Toddler Quality of Life Questionnaire™ (ITQOL) adopts the World Health Organization's definition of health, as a state of complete physical, mental and social wellbeing and not merely the absence of disease. For each concept, item responses are scored, summed, and transformed on a scale from 0 (worst health) to 100 (best health).
Time Frame: Week 0 to 24
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 19 | 17
scores on a scale | 3.4211 (4.8652) | 1.4706 (5.1434)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.08 — Pr(>F) = 0.7846, Nested model using site as a predictor

4. Secondary Outcome: Change in Child Quality of Life as Measured by the Infant Toddler Quality of Life Scale (ITQOL47) - Combined Behavior Scale (CBE) Subscale
Description: he investigators will model child quality of life from Week 0 to Week 24 of the intervention. The Infant Toddler Quality of Life Questionnaire™ (ITQOL) was developed for use in infants and toddlers from 2-months-to-5 years of age. The Infant Toddler Quality of Life Questionnaire™ (ITQOL) adopts the World Health Organization's definition of health, as a state of complete physical, mental and social wellbeing and not merely the absence of disease. For each concept, item responses are scored, summed, and transformed on a scale from 0 (worst health) to 100 (best health).
Time Frame: Week 0 to 24
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 19 | 17
scores on scale | 0.3947 (2.4536) | -0.9804 (2.5939)
Statistical Analysis 1: Comparison: Megestrol; Test type: Superiority; Mean Difference (Final Values) = 0.15 — Pr(>F) = 0.7025, Nested model using site as a predictor

5. Secondary Outcome: Change in Child Quality of Life as Measured by the Child Health Questionnaire Parent Form - CHQ-PF50, 5.1 Behavior (BE) Subscale
Description: Child quality of life in children aged ≥5 years will be assessed using the Child Health Questionnaire Parent Form - CHQ-PF50, a validated parent-reported measure of physical and psychosocial health for children ages 5-18. The CHQ-PF50 contains 50 items assessing 14 health concepts, including physical functioning, emotional/behavioral well-being, social functioning, and family impact.
  The Behavior (BE) subscale evaluates behavioral and emotional adjustment as observed by the parent. Subscale scores range from 0 to 100, with higher scores representing better behavioral health and fewer behavioral problems.
  CHQ-PF50 scores can be analyzed at the subscale level (CHQ Profile Scores) or combined into Summary Scores for physical and psychosocial health. Summary scores are calculated by averaging standardized subscale scores, also ranging from 0 to 100, with higher scores indicating better overall health-related quality of life.
Time Frame: Week 0 to 24
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 10 | 7
scores on a scale | 5.0000 (5.0249) | 8.3333 (6.0059)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.18 — Pr(>F) = 0.6764, Nested model using site as a predictor

6. Secondary Outcome: Change in Child Quality of Life as Measured by the Child Health Questionnaire Parent Form - CHQ-PF50 - 5.2 Global Behavior (GBE) Subscale
Description: Child quality of life in children aged ≥5 years will be assessed using the Child Health Questionnaire Parent Form - CHQ-PF50, a validated parent-reported measure of physical and psychosocial health for children ages 5-18. The CHQ-PF50 includes 50 items covering 14 health concepts, such as physical functioning, emotional/behavioral well-being, social functioning, and family impact.
  The Global Behavior (GBE) subscale assesses overall behavioral and emotional functioning as reported by the parent. Subscale scores range from 0 to 100, with higher scores indicating better global behavioral health and fewer overall behavioral problems.
  CHQ-PF50 scores can be analyzed at the subscale level (CHQ Profile Scores) or combined into Summary Scores for physical and psychosocial health. Summary scores are calculated by averaging standardized subscale scores, also ranging from 0 to 100, with higher scores representing better overall health-related quality of life.
Time Frame: Week 0 to 24
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 10 | 7
scores on a scale | -2.5000 (5.2678) | -0.000000000001 (6.2963)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.09 — Pr(>F) = 0.7649, Nested model using site as a predictor

7. Secondary Outcome: Change in Parent Stress as Measured by the Pediatric Inventory for Parents (PIP36) - Total Frequency Score
Description: The investigators will model parent stress levels from Week 0 to Week 24 of the intervention. The PIP is scored separately for each of the 4 domains (Communication, Emotional Distress, Medical Care, Role Function), across 2 scales: Frequency (F) and Difficulty (D). There is also a total score comprised of the sum for each of the 4 domains, yielding Total F and Total D scores. Items are scored as endorsed by respondents, ranging from 1-5. The range for each of the Total F and Total D scores is 42-210. Higher scores are indicative of worse parent stress outcomes.
Time Frame: Weeks 0 to 24
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 28 | 24
scores on a scale | -20.7500 (5.2481) | -21.2500 (5.6686)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.00 — Pr(>F) = 0.9487, Nested model using site as a predictor

8. Secondary Outcome: Change in Parent Stress as Measured by the Pediatric Inventory for Parents (PIP36) - Total Difficulty Score
Description: as for outcome 7
Time Frame: Weeks 0 to 24
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 28 | 24
scores on a scale | -18.7143 (5.6856) | -21.2083 (6.1411)
Statistical Analysis 1: Comparison: Megestrol; Test type: Superiority; Mean Difference (Final Values) = 0.09 — Pr(>F) = 0.7669, Nested model using site as a predictor

9. Secondary Outcome: Change in Parent Quality of Life as Measured by the SF-36v2 - Emotional Well-Being Subscale
Description: Parent quality of life will be assessed using the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36v2), a widely used, validated self-report measure of general health-related quality of life. The SF-36v2 includes 36 items covering 8 domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health.
  The Emotional Well-Being (Mental Health) subscale measures overall emotional functioning, including mood, anxiety, and psychological distress. Raw subscale scores range from 0 to 100, with higher scores indicating better emotional well-being.
  For analysis, raw subscale scores will be converted to standardized Z-scores, where a Z-score of 0 represents the population mean, and each standard deviation above or below 0 represents deviation from the mean. Higher Z-scores indicate better emotional functioning, while lower Z-scores indicate worse emotional
Time Frame: Week 0 to 24
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 29 | 24
z-score | 0.9655 (2.5131) | 3.0000 (2.7625)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.30 — Pr(>F) = 0.5883, Nested model using site as a predictor

10. Secondary Outcome: Change in Parent Depressive Symptoms Measured by the Patient Health Questionnaire-9 (PHQ-9)
Description: Parent depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated 9-item self-report measure of depression severity based on the 9 criteria for Major Depressive Disorder (MDD) from the DSM. Each item is scored from 0 ("not at all") to 3 ("nearly every day"), yielding a total score ranging from 0 to 27.
  Higher PHQ-9 scores indicate greater severity of depressive symptoms, while lower scores indicate fewer or less severe depressive symptoms. Total score interpretation is commonly as follows: 0-4 = minimal or no depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, 20-27 = severe depression. This measure can be used to assess both the presence of depressive symptoms and changes in symptom severity over time.
Time Frame: Week 0 to 24
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 28 | 23
scores on a scale | -0.5357 (0.9456) | 0.4783 (0.4783)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.52 — Pr(>F) = 0.4749, Nested model using site as a predictor

11. Secondary Outcome: Change in Parent Anxiety Symptoms Measured by the General Anxiety Disorder-7 (GAD-7).
Description: Parent anxiety symptoms will be assessed using the Generalized Anxiety Disorder-7 (GAD-7), a validated 7-item self-report measure that screens for and assesses the severity of common anxiety disorders, including Generalized Anxiety Disorder, Panic Disorder, Social Phobia, and Post-Traumatic Stress Disorder.
  Each item is scored from 0 ("not at all") to 3 ("nearly every day"), yielding a total score range of 0 to 21. Higher scores indicate greater anxiety symptom severity, whereas lower scores indicate fewer or less severe anxiety symptoms.
  Total scores are interpreted as follows: 0-4 = minimal anxiety, 5-9 = mild anxiety, 10-14 = moderate anxiety, 15-21 = severe anxiety. The total GAD-7 score is calculated by summing the scores for all seven items. This measure can be used to assess the presence of clinically significant anxiety symptoms as well as changes in symptom severity over time.
Time Frame: Week 0 to 24
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Megestrol | Placebo
Number analyzed (Participants) | 28 | 23
scores on a scale | -0.9643 (0.7912) | -0.7826 (0.8730)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.02 — Pr(>F) = 0.8781, Nested model using site as a predictor

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Megestrol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 5/36 | 5/34
Other Adverse Events (participants affected / at risk) | 27/36 | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Megestrol (N=36) | Placebo (N=34)
Post-surgical ileus (Gastrointestinal disorders) | 1 (1) | 0
Tachycardia (Cardiac disorders) | 1 (1) | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0
Allergenic reaction to food (Immune system disorders) | 1 (1) | 0
Weight loss (Metabolism and nutrition disorders) | 0 | 1 (1)
Weakness (General disorders) | 0 | 1 (1)
Dehydration (General disorders) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 | 1 (1)
Fever (Infections and infestations) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Megestrol (N=36) | Placebo (N=34)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Ear infection (Infections and infestations) | 3 (5) | 4 (4)
Fever (General disorders) | 8 (10) | 5 (6)
Irritability (Psychiatric disorders) | 2 (2) | 0
Respiratory virus (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 16 (24)
Streptococcal pharyngitis (Infections and infestations) | 2 (2) | 0
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (3)
Weight loss (Metabolism and nutrition disorders) | 2 (3) | 0
High cortisol (Endocrine disorders) | 2 (2) | 0
Low cortisol (Endocrine disorders) | 5 (9) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT03815019/Prot_SAP_000.pdf